CLINICAL TRIAL: NCT04230174
Title: Effect of Ocrelizumab on Neuroinflammation in Multiple Sclerosis as Measured by 11C-PBR28 MR-PET Imaging of Microglia Activation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Caterina Mainero, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019P002865
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine

STUDY DESIGN:
Intervention Model Description: 24 multiple sclerosis patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multiple sclerosis patients (Experimental): Multiple sclerosis patients will be evaluated with 11C-PBR28 MR-PET at baseline before and at 12 month follow up after Ocrelizumab therapy.
  Interventions: Drug: 11C-PBR28

INTERVENTIONS:
Drug: 11C-PBR28 — This study will evaluate, serially, functional and structural tissue changes in the cortex and WM of subjects with RRMS and progressive disease under Ocrelizumab using 11C-PBR28 MR-PET imaging at baseline and at approximately 12-month follow up.

SUMMARY:
Using magnetic resonance-PET (MR-PET) imaging with [11C]PBR28, a second-generation 18kDa translocator protein (TSPO) radiotracer, we have previously demonstrated abnormally high TSPO expression, indicative of microglia activation, across different brain tissue compartments of multiple sclerosis (MS) patients1.

In this study, we propose to study the efficacy of ocrelizumab, a humanized monoclonal antibody that has been shown to decrease neuroinflammation in relapsing-remitting multiple sclerosis (RRMS) and progressive multiple sclerosis (MS) patients.

We will test these effects by studying a cohort of 24 MS patients (12 RRMS, 12 progressive MS). Participants will be studied before (within 3 months prior to initiating treatment) and after treatment with ocrelizumab (~12 month follow up), a therapeutic drug that will be part of their standard medical care. We will use [11C]PBR28 to help determine changes in neuroinflammation.

The purpose of this study is to determine the effects of ocrelizumab treatment on neuroinflammation by analyzing the uptake and distribution of [11C]PBR28 in individuals with multiple sclerosis. The specific aims of the current study are:

1. To assess whether treatment with ocrelizumab in subjects with either relapsing-remitting MS or progressive MS is associated with decreased [11C]PBR28 binding in the cortex and white matter (lesions and normal appearing white matter), suggesting reduced neuroinflammation.
2. To assess whether changes in neuroinflammation under ocrelizumab treatment, as measured by [11C]PBR28 uptake at 12-month follow up relative to baseline, are associated with changes in structural MR metrics of brain tissue damage including white matter lesion load, cortical atrophy, and demyelination in the cortex and in the normal-appearing white matter as measured by magnetization transfer ratio (MTR).
3. To explore whether changes in functional and structural imaging metrics under ocrelizumab are associated with changes in clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. RRMS and/or PMS subtype
3. EDSS between 0 and 7.0
4. Express at least one high-affinity (Ala147) allele of the TSPO receptor for PBR28
5. Initiating Ocrelizumab treatment within the next 3 months

Exclusion Criteria:

1. Hypersensitivity to trial medications
2. History of life-threatening reaction to Ocrelizumab
3. Acute or uncontrolled chronic medical condition
4. Impaired hearing
5. Claustrophobia
6. 300 lbs of greater (weight limit of MRI table)
7. Pregnancy or breastfeeding
8. Sensitivity to imaging agents
9. Contraindications to MRI
10. Use of benzodiazepines, topiramate, doxycycline, mynocicline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Mainero, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 patients signed the consent form.
Pre-assignment Details: Out of the 22 patients that signed the consent form, 2 patients became later ineligible to continue with the baseline study procedures.
Groups:
- Multiple Sclerosis Patients: Multiple sclerosis patients will be evaluated with 11C-PBR28 MR-PET at baseline before and at 12 month follow up after Ocrelizumab therapy.
  This study will evaluate, serially, functional and structural tissue changes in the cortex and brain white matter (lesions and normal appearing white matter) of subjects with RRMS and progressive disease under Ocrelizumab using 11C-PBR28 MR-PET imaging at baseline and at approximately 12-month follow up.
Period: Overall Study
Arm/Group | Multiple Sclerosis Patients
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Patients with multiple sclerosis
Arm/Group | Multiple Sclerosis Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants] — Count of study participants
  Participants
    <=18 years | 0
    Between 18 and 65 years | 20
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at baseline
  years | 43.15 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18
  Black/African American | 1
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: 11C-PBR28 Uptake as Measured by Standardized Uptake Values Normalized by a Pseudoreference Region (SUVR)
Description: The primary endpoint is change in mean 11C-PBR28 SUVR in multiple sclerosis patients after 1-year of ocrelizumab therapy in different brain regions.
Time Frame: Baseline to 12 month
Population: Fifteen MS patients completed the follow-up MR-PET study, which was performed at an average interval of 19.8 days (SD=22.6) after receiving the 1-year ocrelizumab dose. A patient was excluded from the PET analysis after it was discovered that they were using a medication not allowed by the study protocol.
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Multiple sclerosis patients
Number analyzed (Participants) | 14
SUVR
  Baseline SUVR in perilesional white matter | 0.9 (0.19)
  Baseline SUVR in white matter lesions | 0.9 (0.21)
  Baseline SUVR in thalamus | 1.31 (0.26)
  12-month SUVR in perilesional white matter | 0.84 (0.19)
  12-month SUVR in white matter lesions | 0.83 (0.2)
  12-month SUVR in thalamus | 1.23 (0.25)
Statistical Analysis 1: Comparison: Multiple sclerosis patients; Test type: Other — Paired-t test baseline vs follow-up SUVR in white matter lesions of multiple sclerosis patients; p = 0.011, t-test, 2 sided
Statistical Analysis 2: Comparison: Multiple sclerosis patients; Paired-t test baseline vs follow-up SUVR in perilesional white matter multiple sclerosis patients; Test type: Other — Paired-t test; p = 0.018, t-test, 2 sided
Statistical Analysis 3: Comparison: Multiple sclerosis patients; Paired-t test baseline vs follow-up SUVR in the thalamus of multiple sclerosis patients; Test type: Other — Paired-t test; p = 0.047, t-test, 2 sided; A general linear model using the FreeSurfer software was used to assess, vertex-wise, significant paired-wise SUVR differences in post vs pre ocrelizumab treatment in patients across the cortex. A clusterwise correction for multiple comparisons was also applied using a Monte-Carlo simulation with 10,000 iterations (corrected P ≤ 0.05). The surface-based analysis disclosed three clusters of decreased 11C-PBR28 uptake in the right hemisphere (Fig. 4), including insula (p=0.0009), lateral orbitofrontal (p=0.03), and opercular/frontal inferior (p=0.02) areas after adjusting for multiple comparisons

2. Secondary Outcome: Magnetization Transfer Ratio (MTR)
Description: Secondary endpoint is changes in mean magnetization transfer ratio (MTR) in cortex and normal appearing white matter (NAWM) of multiple sclerosis patients after 1-year of ocrelizumab therapy. MTR is defined as: S0 - S_MT/S0; where S0 is the signal intensity without the magnetization transfer (MT) pulse and S_MT is the signal intensity with the MT pulse. It is dimensionless because it is defined as a ratio of two signals with the same physical units, so the units cancel out. Larger MTR indicate stronger interaction between free water protons and macromolecular-bound protons.
Time Frame: Baseline to 12-month
Population: Longitudinal MTR scans were acquired in 15 patients; in one subject, however, the MT_off acquisition was not completed due to early scan termination as the subject was unable to tolerate the scan duration. MTR maps from another subject were excluded from the group analysis due to severe motion artifacts.
Measure: Mean (Standard Deviation); unit: % of MTR
Arm/Group | Multiple sclerosis patients
Number analyzed (Participants) | 13
% of MTR
  Baseline NAWM MTR | 27.9 (1.4)
  Baseline cortical MTR | 17.3 (0.9)
  12-month NAWM MTR | 27.0 (1.9)
  12-month cortical MTR | 16.8 (1.1)
Statistical Analysis 1: Comparison: Multiple sclerosis patients; Baseline vs follow-up MTR in NAWM; Test type: Other — Paired-t test; p = 0.07, t-test, 2 sided
Statistical Analysis 2: Comparison: Multiple sclerosis patients; Baseline vs follow-up MTR in cortex; Test type: Other — Paired-t test; p = 0.024, t-test, 2 sided

3. Secondary Outcome: Cortical Thickness
Description: Secondary endpoint is changes in cortical thickness after 1-year ocrelizumab treatment in patients with multiple sclerosis.
Time Frame: Baseline to 12-month
Population: A patient was excluded from the study analysis after it was discovered that they were using a medication not allowed by the study protocol.
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | Multiple sclerosis patients
Number analyzed (Participants) | 14
mm2
  Baseline cortical thickness | 2.35 (0.09)
  12-month cortical thickness | 2.35 (0.07)
Statistical Analysis 1: Comparison: Multiple sclerosis patients; Changes in cortical thickness after 1-year ocrelizumab treatment in patients with multiple sclerosis; Test type: Other — Paired-t test; p = 0.69, t-test, 2 sided

4. Secondary Outcome: White Matter (WM) Lesion Volume
Description: Secondary endpoint is changes in WM lesion load after 1-year of ocrelizumab therapy in patients with MS.
Time Frame: Baseline to 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm cubic
Arm/Group | Multiple sclerosis patients
Number analyzed (Participants) | 14
mm cubic
  Baseline white matter lesion volume | 6248 (7314)
  12-month white matter lesion volume | 6021 (6821)
Statistical Analysis 1: Comparison: Multiple sclerosis patients; Wilcoxon related samples test comparing baseline vs follow-up changes in white matter lesion volume of multiple sclerosis patients; Test type: Other — Wilcoxon related samples test; p = 0.64, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The study period during which all AE are reported begins after informed consent is obtained and initiation of study treatment and ends 30 days following the last administration of radiotracer and MR-PET or study discontinuation/termination, whichever is earlier, approximately up to 14-15 months.
Arm/Group | Multiple Sclerosis Patients
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Sclerosis Patients (N=20)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Bronchopneumonia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Sclerosis Patients (N=20)
Covid-19 (Infections and infestations) | 4 (4)
Typical multiple sclerosis relapse (Nervous system disorders) | 2 (2)
Urinary infection (Infections and infestations) | 1 (1)
Hiatal hernia (Gastrointestinal disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ocrevus infusion reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT04230174/Prot_SAP_001.pdf